CLINICAL TRIAL: NCT02080871
Title: Evaluation of the Gore(R) Viabahn(R) Balloon Expandable Endoprosthesis (VIABAHN BX) for the Treatment of Occlusive Disease in the Common and External Iliac Arteries.
Brief Title: A Study of the Gore VIABAHN BX for Treatment of Occlusive Disease in the Iliac Arteries.
Acronym: VBXFLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BES 10-07
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-12

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; Stent; Claudication; Viabahn; Gore; Endoprosthesis; Vascular Diseases; Cardiovascular Diseases; Iliac Occlusive Disease; Balloon Expandable; Stent-graft; VBX
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Gore VIABAHN BX (Experimental): Balloon expandable stenting of iliac occlusive disease
  Interventions: Device: Stenting of the Common and/or External Iliac Arteries

INTERVENTIONS:
Device: Stenting of the Common and/or External Iliac Arteries — Balloon expandable stenting of iliac occlusive disease.

SUMMARY:
Evaluation of the Gore(R) VIABAHN BX for the treatment of arterial occlusive disease in the common and/or external iliac arteries.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, non-randomized single-arm clinical study to evaluate the safety and efficacy of the VIABAHN BX for the treatment of arterial occlusive disease in patients with de novo or restenotic lesions in the common and/or external iliac arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old;
2. Patient is male, infertile female, or female of childbearing potential practicing an acceptable method of preventing pregnancy;
3. Patient or legal representative is willing to give written informed consent;
4. Patient is capable of complying with protocol requirements, including all follow-up visits;
5. Patient has symptomatic claudication or rest pain without tissue loss (Rutherford Categories 2-4).
6. Patient has de novo or restenotic target lesion(s) in the common and/or external iliac artery;
7. Patient has one or more regions of stenosis ≥ 50% in the target vessel, based on visual estimate;
8. Patient has a target vessel diameter visually estimated to be approximately between 5 mm and 13 mm;
9. Patient has adequate ipsilateral blood flow including at least one sufficient (<50% stenotic) infrapopliteal run-off vessel not requiring intervention (per side to be intervened on).
10. Patient has a total target lesion length visually estimated to be ≤110 mm which can be treated with a maximum of three VIABAHN BX endoprostheses;
11. Patient has no more than two discrete ipsilateral lesions that can be treated with no more than three VIABAHN BX endoprostheses [OR] Patient has bilateral disease consisting of only one target lesion per side that can be treated with no more than a total of three VIABAHN BX endoprostheses;
12. Patient has the device advanced across the target lesion(s) and positioned for deployment.

Exclusion Criteria:

1. Patient has a life expectancy of less than 1 year;
2. Patient has a known allergy to stent graft components, including stainless steel or heparin;
3. Patient has a known intolerance to antiplatelet, anticoagulant, or thrombolytic medications that would prevent compliance with the protocol;
4. Patient has a condition (unrelated to the study) that is expected to require indefinite, or lifelong, anticoagulation
5. Patient has an uncorrected bleeding disorder (platelet count < 80,000/µL);
6. Patient has severe chronic renal insufficiency (serum creatinine level > 2.5mg/dL) and not on hemodialysis;
7. Patient has a known hypercoagulability that cannot be corrected;
8. Patient has evidence of a blood borne infection;
9. Patient has had vascular access/catheterization in the lower extremity within 30 days of study enrollment;
10. Patient has had a previous or planned coronary intervention within 30 days prior to enrollment in this study or required at time of study procedure;
11. Patient has had a previous or planned bypass surgery in the target leg, or a bypass that occurs at the time of the index procedure;
12. Patient is currently participating in this or another investigative clinical study.
13. Patient has a stent or stent graft located within or immediately adjacent (≤5mm) to study lesion(s);
14. Patient has evidence of angiographically visible thrombus within or adjacent to the target lesion(s);
15. Patient has aneurysmal dilation proximal or distal to the target lesion(s) that would interfere with the placement of the device;
16. Patient has a target lesion requiring atherectomy or any ablative device to facilitate stent delivery;
17. Patient has a target lesion situated in such a way that an implanted device will prevent blood flow or perfusion to the internal iliac artery if patent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bismuth, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (27):
- United States (26):
  - St. Luke's Medical Center, Phoenix, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Coastal Vascular Institute, Pensacola, Florida
  - Cardiovascular Associates, Elk Grove Village, Illinois
  - Iowa Methodist Medical Center, West Des Moines, Iowa
  - University of Louisville, Louisville, Kentucky
  - Essentia Institute for Rural Health / St Mary's Hospital, Duluth, Minnesota
  - North Memorial Heart & Vascular Institute, Plymouth, Minnesota
  - Advanced Vascular Associates, Morristown, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Research Foundation SUNY Buffalo, Buffalo, New York
  - Cornell University, New York, New York
  - Sanford Clinic - Clinical Research, Fargo, North Dakota
  - Ohio Health, Columbus, Ohio
  - Holy Spirit Cardiovascular Institute, Camp Hill, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - MUSC, Charleston, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - University Surgical Associates, Chattanooga, Tennessee
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - The Methodist Hospital, Houston, Texas
  - Sentara Medical Group, Norfolk, Virginia
- Auckland City Hospital, Auckland, New Zealand

REFERENCES:
- [Derived] Holden A, Takele E, Hill A, Sakhuja R, Metzger C, Gray BH, Cavadino A. Long-Term Follow-up of Subjects With Iliac Occlusive Disease Treated With the Viabahn VBX Balloon-Expandable Endoprosthesis. J Endovasc Ther. 2025 Feb;32(1):68-76. doi: 10.1177/15266028231165723. Epub 2023 Apr 19. PMID 37073512
- [Derived] Panneton JM, Bismuth J, Gray BH, Holden A. Three-Year Follow-up of Patients With Iliac Occlusive Disease Treated With the Viabahn Balloon- Expandable Endoprosthesis. J Endovasc Ther. 2020 Oct;27(5):728-736. doi: 10.1177/1526602820920569. Epub 2020 Apr 24. PMID 32329658
- [Derived] Bismuth J, Gray BH, Holden A, Metzger C, Panneton J; VBX FLEX Study Investigators. Pivotal Study of a Next-Generation Balloon-Expandable Stent-Graft for Treatment of Iliac Occlusive Disease. J Endovasc Ther. 2017 Oct;24(5):629-637. doi: 10.1177/1526602817720463. Epub 2017 Jul 12. PMID 28697693

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gore VIABAHN BX
Started | 134
Completed (Completion of the primary outcome measure (9 months). The study is in long term follow-up.) | 132
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Iliac Stenting: Balloon expandable stenting of iliac occlusive disease
  Stenting of the Common and/or External Iliac Arteries: Balloon expandable stenting of iliac occlusive disease.
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] — Adults >/= 18 years
  years | 66 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 128
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 122
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 27
  United States | 107

OUTCOME MEASURES:

1. Primary Outcome: Composite of Major Adverse Events (MAEs)
Description: Percentage of study subjects experiencing a major adverse event (MAE) defined as: device or procedure-related death within 30 days, myocardial infarction (MI) within 30 days, target lesion revascularization (TLR) within 9 months or major amputation of the target limb within 9 months.
Time Frame: 9 months
Population: Population includes enrolled subjects who either experienced the defined event or were followed for at least 240 days.
Measure: Number (95% Confidence Interval); unit: percentage of subjects experiencing MAE
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 132
percentage of subjects experiencing MAE | 2.3 [0.5 to 6.5]
Statistical Analysis 1: Comparison: Iliac Stenting; The sample size obtains over 90% power to statistically show the probability that a subject will experience an MAE with use of the study device is less than 17% when 12% or less of the subjects are lost to follow up prior to 9 months; Test type: Other — This was a single-arm study designed to compare the primary outcome result to a performance goal based on published literature. The null hypothesis was the probability of a subject experiencing a Major Adverse Event (MAE) with use of study device is at least 17%. The alternate hypothesis was the probability of a subject experiencing a Major Adverse Event (MAE) with use of the study device is less than 17%; p < 0.001, one-sided binomial exact test

2. Secondary Outcome: Acute Procedural Success
Description: Number of subjects who experienced Acute Procedural Success defined as less than or equal to 30% residual stenosis prior to procedure completion and no device- or procedure-related SAEs before discharge.
Time Frame: Discharge
Population: Population includes subjects followed through discharge and had relevant procedural data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Participants | 130

3. Secondary Outcome: 30-Day Clinical Success
Description: Number of subjects who experienced 30-Day Clinical Success defined as an improvement of at least one Rutherford Category at the 30-day visit as compared to pre-procedure and no device- or procedure-related SAEs within 30 days of the index procedure.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 119
Participants | 108

4. Secondary Outcome: Percentage of Participants With Primary Patency
Description: Kaplan-Meier estimate of primary patency at 30 days.
Time Frame: 30 Days
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: survival percentage by subject
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
survival percentage by subject | 99.2 [94.8 to 99.9]

5. Secondary Outcome: Percentage of Participants With Primary Patency
Description: Kaplan-Meier estimate of primary patency at 9 months.
Time Frame: 9 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: survival percentage by subject
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
survival percentage by subject | 96.7 [91.5 to 98.8]

6. Secondary Outcome: Percentage of Participants With Primary Assisted Patency
Description: Kaplan-Meier estimate of primary assisted patency at 30 days.
Time Frame: 30 Days
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: survival percentage by subject
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
survival percentage by subject | 99.2 [94.8 to 99.9]

7. Secondary Outcome: Percentage of Participants With Primary Assisted Patency
Description: Kaplan-Meier estimate of primary assisted patency at 9 months.
Time Frame: 9 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: survival percentage by subject
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
survival percentage by subject | 99.2 [94.8 to 99.9]

8. Secondary Outcome: Percentage of Participants With Secondary Patency
Description: Kaplan-Meier estimate of secondary patency at 30 days.
Time Frame: 30 Days
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: survival percentage by subject
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
survival percentage by subject | 99.2 [94.8 to 99.99]

9. Secondary Outcome: Percentage of Participants With Secondary Patency
Description: Kaplan-Meier estimate of secondary patency at 9 months.
Time Frame: 9 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: survival percentage by subject
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
survival percentage by subject | 99.2 [94.8 to 99.9]

10. Secondary Outcome: Percentage of Participants With Freedom From Target Lesion Revascularization (TLR)
Description: Kaplan-Meier estimate of freedom from target lesion revascularization (TLR) at 30 days.
Time Frame: 30 Days
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 100 [100 to 100]

11. Secondary Outcome: Percentage of Participants With Freedom From Target Lesion Revascularization (TLR)
Description: Kaplan-Meier estimate of freedom from target lesion revascularization (TLR) at 9 months.
Time Frame: 9 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 97.7 [92.9 to 99.2]

12. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Lesion Revascularization (CD-TLR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target lesion revascularization (CD-TLR) at 30 days.
Time Frame: 30 Days
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 100 [100 to 100]

13. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Lesion Revascularization (CD-TLR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target lesion revascularization (CD-TLR) at 9 months.
Time Frame: 9 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 98.4 [93.8 to 99.6]

14. Secondary Outcome: Percentage of Participants With Freedom From Target Vessel Revascularization (TVR)
Description: Kaplan-Meier estimate of freedom from target vessel revascularization (TVR) at 30 days.
Time Frame: 30 Days
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 100 [100 to 100]

15. Secondary Outcome: Percentage of Participants With Freedom From Target Vessel Revascularization (TVR)
Description: Kaplan-Meier estimate of freedom from target vessel revascularization (TVR) at 9 months.
Time Frame: 9 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 97.7 [92.9 to 99.2]

16. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Vessel Revascularization (CD-TVR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target vessel revascularization (CD-TVR) at 30 days.
Time Frame: 30 Days
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 100 [100 to 100]

17. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Vessel Revascularization (CD-TVR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target vessel revascularization (CD-TVR) at 9 months
Time Frame: 9 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 97.7 [92.9 to 99.2]

18. Secondary Outcome: Number of Participants With Change in Rutherford Category
Description: Number of participants with change in Rutherford Category from pre-procedure at 30 days.
  Rutherford Categories:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 30 Days
Population: Population includes subjects followed for at least 23 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 118
Participants
  Improved Rutherford Category | 111
  Maintained Rutherford Category | 6
  Worsened Rutherford Category | 1

19. Secondary Outcome: Number of Participants With Change in Rutherford Category
Description: Number of participants with change in Rutherford Category from pre-procedure at 9 months.
  Rutherford Categories:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days and relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 112
Participants
  Improved Rutherford Category | 106
  Maintained Rutherford Category | 6
  Worsened Rutherford Category | 0

20. Secondary Outcome: Change in Ankle Brachial Index (ABI)
Description: Ankle brachial Index (ABI) is a common assessment of peripheral artery disease (PAD) and is obtained by comparing the systolic blood pressure of the legs to the systolic blood pressure of the arms. A normal resting ABI is .9 to 1.3. A resting ABI of less than .9 is abnormal. An outcome of a mean ABI above .9 and below 1.3 is considered a success.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 23 days and had relevant data.
Measure: Mean (Full Range); unit: ratio index
Units Other Than Participants: limbs
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 117
Number analyzed (limbs) | 174
ratio index | .97 [.42 to 1.34]

21. Secondary Outcome: Change in Ankle Brachial Index (ABI)
Description: as for outcome 20
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days and had relevant data.
Measure: Mean (Full Range); unit: ratio index
Units Other Than Participants: limbs
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 111
Number analyzed (limbs) | 169
ratio index | 0.97 [.42 to 1.43]

22. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Mobility
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Mobility) from pre-procedure at 30 days.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 23 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 51
  Maintained | 57
  Worsened | 7

23. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Mobility
Description: Patient reported outcome based on study questionnaire. Number of participants with change in Functional Status (EQ5D - Mobility) from pre-procedure at 9 months.
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 114
Participants
  Improved | 48
  Maintained | 62
  Worsened | 4

24. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Self Care
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Self Care) from pre-procedure at 30 days.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 5
  Maintained | 108
  Worsened | 2

25. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Self Care
Description: Patient reported outcome based on study questionnaire. Number of participants with change in Functional Status (EQ5D - Self Care) from pre-procedure at 9 months.
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 114
Participants
  Improved | 6
  Maintained | 105
  Worsened | 3

26. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Usual Activities
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Usual Activities) from pre-procedure at 30 days.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 52
  Maintained | 55
  Worsened | 8

27. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Usual Activities
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Usual Activities) from pre-procedure at 9 months.
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 114
Participants
  Improved | 53
  Maintained | 57
  Worsened | 4

28. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Pain/Discomfort
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Pain/Discomfort) from pre-procedure at 30 days.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 56
  Maintained | 49
  Worsened | 10

29. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Pain/Discomfort
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Pain/Discomfort) from pre-procedure at 9 months.
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 114
Participants
  Improved | 49
  Maintained | 55
  Worsened | 10

30. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Anxiety/Depression
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Anxiety/Depression) from pre-procedure at 30 days.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 27
  Maintained | 82
  Worsened | 6

31. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Anxiety/Depression
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Anxiety/Depression) from pre-procedure at 9 months.
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 114
Participants
  Improved | 28
  Maintained | 79
  Worsened | 7

32. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Own Health State
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Own Health State) from pre-procedure at 30 days.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 114
Participants
  Improved | 22
  Maintained | 84
  Worsened | 8

33. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Own Health State
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Own Health State) from pre-procedure at 9 months.
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 113
Participants
  Improved | 23
  Maintained | 73
  Worsened | 17

34. Secondary Outcome: Number of Participants With Improvement in Functional Status at 30 Days - Walking Improvement Questionnaire (WIQ)
Description: Patient reported outcome based on study questionnaire. Percentage of subjects with improvement on WIQ from pre-procedure at 30 days.
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants | 106

35. Secondary Outcome: Number of Participants With Improvement in Functional Status 9 Months - Walking Improvement Questionnaire (WIQ)
Description: Patient reported outcome based on study questionnaire. Percentage of subjects with improvement on WIQ from pre-procedure at 9 months.
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days and had relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 114
Participants | 102

36. Secondary Outcome: Percentage of Participants With Primary Patency
Description: Kaplan-Meier estimate of primary patency at 12 months.
Time Frame: 12 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: survival percentage by subject
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
survival percentage by subject | 94.4 [88.7 to 97.3]

37. Secondary Outcome: Percentage of Participants With Primary Assisted Patency
Description: Kaplan-Meier estimate of primary assisted patency at 12 months.
Time Frame: 12 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: survival percentage by subject
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
survival percentage by subject | 98.4 [93.9 to 99.6]

38. Secondary Outcome: Percentage of Participants With Secondary Patency
Description: Kaplan-Meier estimate of secondary patency at 12 months.
Time Frame: 12 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: survival percentage by subject
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
survival percentage by subject | 99.2 [94.8 to 99.6]

39. Secondary Outcome: Percentage of Participants With Freedom From Target Lesion Revascularization (TLR)
Description: Kaplan-Meier estimate of freedom from target lesion revascularization (TLR) at 12 months.
Time Frame: 12 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 95.4 [90.1 to 97.9]

40. Secondary Outcome: Percentage of Participants With Freedom From Target Lesion Revascularization (TLR)
Description: Kaplan-Meier estimate of freedom from target lesion revascularization (TLR) at 24 months.
Time Frame: 24 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 93.1 [87.1 to 96.3]

41. Secondary Outcome: Percentage of Participants With Freedom From Target Lesion Revascularization (TLR)
Description: Kaplan-Meier estimate of freedom from target lesion revascularization (TLR) at 36 months.
Time Frame: 36 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 91.4 [84.9 to 95.1]

42. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Lesion Revascularization (CD-TLR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target lesion revascularization (CD-TLR) at 12 months.
Time Frame: 12 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 97.7 [93.1 to 99.3]

43. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Lesion Revascularization (CD-TLR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target lesion revascularization (CD-TLR) at 24 months.
Time Frame: 24 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 97.7 [93.1 to 99.3]

44. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Lesion Revascularization (CD-TLR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target lesion revascularization (CD-TLR) at 36 months.
Time Frame: 36 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 97.7 [93.1 to 99.3]

45. Secondary Outcome: Percentage of Participants With Freedom From Target Vessel Revascularization (TVR)
Description: Kaplan-Meier estimate of freedom from target vessel revascularization (TVR) at 12 months.
Time Frame: 12 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 95.4 [90.1 to 97.9]

46. Secondary Outcome: Percentage of Participants With Freedom From Target Vessel Revascularization (TVR)
Description: Kaplan-Meier estimate of freedom from target vessel revascularization (TVR) at 24 months.
Time Frame: 24 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 92.3 [86.1 to 95.8]

47. Secondary Outcome: Percentage of Participants With Freedom From Target Vessel Revascularization (TVR)
Description: Kaplan-Meier estimate of freedom from target vessel revascularization (TVR) at 36 months.
Time Frame: 36 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 90.6 [84.0 to 94.5]

48. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Vessel Revascularization (CD-TVR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target vessel revascularization (CD-TVR) at 12 months
Time Frame: 12 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 97.7 [93.1 to 99.3]

49. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Vessel Revascularization (CD-TVR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target vessel revascularization (CD-TVR) at 24 months
Time Frame: 24 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 96.9 [92.0 to 98.8]

50. Secondary Outcome: Percentage of Participants With Freedom From Clinically-Driven Target Vessel Revascularization (CD-TVR)
Description: Kaplan-Meier estimate of freedom from clinically-driven target vessel revascularization (CD-TVR) at 36 months
Time Frame: 36 Months
Population: Population includes all subjects meeting eligibility.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 134
Percentage of participants | 96.1 [90.9 to 98.4]

51. Secondary Outcome: Number of Participants With Change in Rutherford Category
Description: Number of participants with change in Rutherford Category from pre-procedure at 12 months.
  Rutherford Categories:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 12 Months
Population: Population includes subjects available at 12 Months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 114
Participants
  Improved Rutherford Category | 108
  Maintained Rutherford Category | 6
  Worsened Rutherford Category | 0

52. Secondary Outcome: Number of Participants With Change in Rutherford Category
Description: Number of participants with change in Rutherford Category from pre-procedure at 24 months.
  Rutherford Categories:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 24 Months
Population: Population includes subjects available at 24 Months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 102
Participants
  Improved Rutherford Category | 96
  Maintained Rutherford Category | 5
  Worsened Rutherford Category | 1

53. Secondary Outcome: Number of Participants With Change in Rutherford Category
Description: Number of participants with change in Rutherford Category from pre-procedure at 36 months.
  Rutherford Categories:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 36 Months
Population: Population includes subjects available at 36 Months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 89
Participants
  Improved Rutherford Category | 82
  Maintained Rutherford Category | 7
  Worsened Rutherford Category | 0

54. Secondary Outcome: Change in Ankle Brachial Index (ABI)
Description: as for outcome 20
Time Frame: 12 Months
Population: Population includes subjects available at 12 Months with relevant data.
Measure: Mean (Full Range); unit: ratio index
Units Other Than Participants: Limbs
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 120
Number analyzed (Limbs) | 165
ratio index | 0.19 [-.90 to .82]

55. Secondary Outcome: Change in Ankle Brachial Index (ABI)
Description: as for outcome 20
Time Frame: 24 Months
Population: Population includes subjects available at 24 Months with relevant data.
Measure: Mean (Full Range); unit: ratio index
Units Other Than Participants: Limbs
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 117
Number analyzed (Limbs) | 148
ratio index | .17 [-1.0 to 0.79]

56. Secondary Outcome: Change in Ankle Brachial Index (ABI)
Description: as for outcome 20
Time Frame: 36 Months
Population: Population includes subjects available at 36 Months with relevant data.
Measure: Mean (Full Range); unit: ratio index
Units Other Than Participants: Limbs
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 102
Number analyzed (Limbs) | 123
ratio index | 0.17 [-0.40 to 0.75]

57. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Mobility
Description: Patient reported outcome based on study questionnaire. Number of participants with change in Functional Status (EQ5D - Mobility) from pre-procedure at 12 months.
Time Frame: 12 Months
Population: Population includes subjects available at 12 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 44
  Maintained | 66
  Worsened | 5

58. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Mobility
Description: Patient reported outcome based on study questionnaire. Number of participants with change in Functional Status (EQ5D - Mobility) from pre-procedure at 24 months.
Time Frame: 24 Months
Population: Population includes subjects available at 24 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 103
Participants
  Improved | 45
  Maintained | 53
  Worsened | 5

59. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Mobility
Description: Patient reported outcome based on study questionnaire. Number of participants with change in Functional Status (EQ5D - Mobility) from pre-procedure at 36 months.
Time Frame: 36 Months
Population: Population includes subjects available at 36 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 90
Participants
  Improved | 43
  Maintained | 43
  Worsened | 4

60. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Self Care
Description: Patient reported outcome based on study questionnaire. Number of participants with change in Functional Status (EQ5D - Self Care) from pre-procedure at 12 months.
Time Frame: 12 Months
Population: Population includes subjects available at 12 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 6
  Maintained | 106
  Worsened | 3

61. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Self Care
Description: Patient reported outcome based on study questionnaire. Number of participants with change in Functional Status (EQ5D - Self Care) from pre-procedure at 24 months.
Time Frame: 24 Months
Population: Population includes subjects available at 24 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 103
Participants
  Improved | 5
  Maintained | 93
  Worsened | 5

62. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Self Care
Description: Patient reported outcome based on study questionnaire. Number of participants with change in Functional Status (EQ5D - Self Care) from pre-procedure at 36 months.
Time Frame: 36 Months
Population: Population includes subjects available at 36 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 90
Participants
  Improved | 4
  Maintained | 84
  Worsened | 2

63. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Usual Activities
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Usual Activities) from pre-procedure at 12 months.
Time Frame: 12 Months
Population: Population includes subjects available at 12 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 51
  Maintained | 55
  Worsened | 9

64. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Usual Activities
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Usual Activities) from pre-procedure at 24 months.
Time Frame: 24 Months
Population: Population includes subjects available at 24 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 103
Participants
  Improved | 44
  Maintained | 51
  Worsened | 8

65. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Usual Activities
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Usual Activities) from pre-procedure at 36 months.
Time Frame: 36 Months
Population: Population includes subjects available at 36 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 90
Participants
  Improved | 44
  Maintained | 42
  Worsened | 4

66. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Pain/Discomfort
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Pain/Discomfort) from pre-procedure at 12 months.
Time Frame: 12 Months
Population: Population includes subjects available at 12 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 59
  Maintained | 44
  Worsened | 12

67. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Pain/Discomfort
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Pain/Discomfort) from pre-procedure at 24 months.
Time Frame: 24 Months
Population: Population includes subjects available at 24 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 103
Participants
  Improved | 49
  Maintained | 41
  Worsened | 13

68. Other Pre Specified Outcome: Device or Procedure-related Death
Description: Number of subjects experiencing a device or procedure-related death within 30 Days - Component of primary outcome
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 133
Participants | 0

69. Other Pre Specified Outcome: Myocardial Infarction (MI)
Description: Number of subjects experiencing a myocardial infarction (MI) within 30 Days - Component of primary outcome
Time Frame: 30 Days
Population: Population includes subjects followed for at least 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 133
Participants | 0

70. Other Pre Specified Outcome: Target Lesion Revascularization (TLR)
Description: Number of subjects experiencing a target lesion revascularization (TLR) within 9 months - Component of primary outcome
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 132
Participants | 3

71. Other Pre Specified Outcome: Major Amputation
Description: Number of subjects experiencing a major amputation of the target limb within 9 months - Component of primary outcome
Time Frame: 9 Months
Population: Population includes subjects followed for at least 240 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 132
Participants | 0

72. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Pain/Discomfort
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Pain/Discomfort) from pre-procedure at 36 months.
Time Frame: 36 Months
Population: Population includes subjects available at 36 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 90
Participants
  Improved | 39
  Maintained | 44
  Worsened | 7

73. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Anxiety/Depression
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Anxiety/Depression) from pre-procedure at 12 months.
Time Frame: 12 Months
Population: Population includes subjects available at 12 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 115
Participants
  Improved | 25
  Maintained | 82
  Worsened | 8

74. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Anxiety/Depression
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Anxiety/Depression) from pre-procedure at 24 months.
Time Frame: 24 Months
Population: Population includes subjects available at 24 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 103
Participants
  Improved | 25
  Maintained | 71
  Worsened | 7

75. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Anxiety/Depression
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Anxiety/Depression) from pre-procedure at 36 months.
Time Frame: 36 Months
Population: Population includes subjects available at 36 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 90
Participants
  Improved | 27
  Maintained | 58
  Worsened | 5

76. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Own Health State
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Own Health State) from pre-procedure at 12 months.
Time Frame: 12 Months
Population: Population includes subjects available at 12 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 114
Participants
  Improved | 23
  Maintained | 77
  Worsened | 14

77. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Own Health State
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Own Health State) from pre-procedure at 24 months.
Time Frame: 24 Months
Population: Population includes subjects available at 24 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 101
Participants
  Improved | 19
  Maintained | 69
  Worsened | 13

78. Secondary Outcome: Number of Participants With Change in Functional Status - EQ5D - Own Health State
Description: Patient reported outcome based on study questionnaire. Number of participants with change in functional status (EQ5D - Own Health State) from pre-procedure at 36 months.
Time Frame: 36 Months
Population: Population includes subjects available at 36 months with relevant data.
Measure: Count of Participants; unit: Participants
Arm/Group | Iliac Stenting
Number analyzed (Participants) | 89
Participants
  Improved | 21
  Maintained | 56
  Worsened | 12

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Iliac Stenting
All-Cause Mortality (participants affected / at risk) | 1/134
Serious Adverse Events (participants affected / at risk) | 30/134
Other Adverse Events (participants affected / at risk) | 0/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iliac Stenting (N=134)
Hemorrhagic anemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Congestive cardiac failure aggravated (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Chest pain (non-cardiac) (General disorders) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Surgical wound infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (1)
Dislocation of ankle (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hematoma (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Cancer of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Vascular dementia (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Claudication (Vascular disorders) | 2 (3)
Femoral artery dissection (Vascular disorders) | 1 (1)
Groin hematoma (Vascular disorders) | 1 (1)
Hypovolemic shock (Vascular disorders) | 1 (1)
Leg ischemia (Vascular disorders) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease aggravated (Vascular disorders) | 1 (1)
Poor peripheral perfusion (Vascular disorders) | 1 (1)
Superficial femoral arterial stenosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No